CLINICAL TRIAL: NCT01147263
Title: Prevalence and Mechanism of Palpitations and Tachycardia in Fibromyalgia Syndrome
Brief Title: Palpitations and Tachycardia in Fibromyalgia Syndrome
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Jacob N Ablin MD, Tel Aviv Sourasky medical center
Other Study IDs: TASMC-10-JA-0678-09-CTIL
Record Dates: First submitted 2010-06-17; First posted 2010-06-22 (Estimated); Last update posted 2010-06-22 (Estimated); Status verified 2010-06

CONDITIONS: Fibromyalgia Syndrome
Keywords: Fibromyalgia; Autonomic dysfunction; Tachycardia; Palpitations
MeSH Terms: conditions — Fibromyalgia; Primary Dysautonomias; Tachycardia

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients diagnosed with Fibromyalgia
  Interventions: Other: Evaluation of autonomic parameters

INTERVENTIONS:
Other: Evaluation of autonomic parameters — Physical examination, ECG, Loop recorder, Heart rate variability evaluation

SUMMARY:
Clinically Characterized by the presence of chronic widespread pan and tenderness, Fibromyalgia (FM) is one of the most common "functional" syndromes. FM is currently conceived of as representing a prototype of central pain, i.e. a condition in which sensitization of the central nervous system results in a overall increase in the processing of painful stimuli, as well as an impairment of pain inhibition. This condition is responsible for significant a social and economic burden and is estimated to affect up to 5% of all women. The 1990 American College of Rheumatology (ACR) classification criteria for FM are the current standard for studying FM, and require the presence of widespread pain lasting over 3 months, as well as documentation of tenderness in at least 11 of 18 pre-defined "tender points. Multiple additional symptoms, which are not part of the classification criteria, include among others sleep disturbances, mood disturbances, cognitive dysfunction, vulvodynia, dysmenorrhea, sexual dysfunction and weight fluctuations. In addition, FM is well known to overlap both clinically and epidemiologically with an ever increasing number of other "functional" disorders, including irritable bowel syndrome (IBS), Temporomandibular joint disorder (TMJD), functional dyspepsia etc. In addition to the central symptom of pain, FM patients frequently complain of non- specific symptoms which are potentially autonomically - mediated. Thus, palpitations, fatigue and inability to stand for long periods of time are all common complaints. About 80-90 percent of FM patients have one or more symptoms associated with autonomic dysfunction. The most common of them is presyncope (62.5%), followed by syncope (12.5%), palpitations on standing (12.5%) and dizziness (12.5%) (14). Some of these symptoms overlap with those of the postural tachycardia syndrome (POTS). POTS is a common dysautonomia, characterized by remarkable increased heart rate during the assumption of the upright posture (>30 bpm). According to our experience, FM is found, at least, in 15% of POTS patients. But, no data exists about the incidence of POTS in patients with FM.The role of the autonomic nervous system (ANS) in initiating and maintaining the syndrome of FM has been studies (and debated) over the last decade. The ANS is an extremely complex system, regulating involuntary body functions, including heart rate, intestinal motility, urination, and sexual activity, among many other variables. Notably, the vagus has an inhibitory effect on pain. Deterioration in the vagal control is "associated" with increased pain sensation. Previous studies have indicated that FM patients may have an increase in sympathetic control over the cardiovascular system with a reciprocal decrease in parasympathetic control. High sympathetic tone is usually associated with a lower threshold to pain. But, the contribution of the ANS to the pathogenesis of FM syndrome remains unclear. Evidently, the ANS interacts with other components of the CNS in the pathogenesis of FM, including pain processing centers in the thalamus and amygdala, as well as with the hypothalamic-pituitary-adrenal (HPA) axis.

ELIGIBILITY:
Inclusion Criteria:

* ACR 1990 criteria for fibromyalgia: widespread pain lasting 3 months
* Tenderness in 11 of 18 points

Exclusion Criteria:

* Unable to provide informed concent
* Known tachyarrhythmia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Consecutive patients attending a fibromyalgia clinic, fullfilling ACR 1990 criteria for classification of fibromyalgia
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2010-07; Primary Completion 2011-06 (Estimated); Study Completion 2012-06 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Tel Aviv Sourasky medical center, Tel Aviv, Israel